CLINICAL TRIAL: NCT01674790
Title: Exploring Potential Synergistic Effects of Aerobic Exercise and Cognitive Training on Cognition After Stroke.
Brief Title: Combined Effects of Aerobic Exercise and Cognitive Training on Cognition After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marilyn MacKay-Lyons (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government); Dalhousie University (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor-Investigator, Marilyn MacKay-Lyons, Affiliated Scientist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Priming Study
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cognitive Training; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AEROBIC group (Experimental): 6-week program of one 20-min session of aerobic training and one 20-min session of ROM exercise 5 days/week.
  Interventions: Behavioral: Aerobic training; Behavioral: Range of motion exercise
- COGNITIVE group (Experimental): 6-week program of one 20-min session of cognitive training and one 20-min session of ROM exercise 5 days/week.
  Interventions: Behavioral: Cognitive training; Behavioral: Range of motion exercise
- AEROBIC + COGNITIVE group (Experimental): 6-week program of one 20-min session of aerobic training and one 20-min session of cognitive training 5 days/week.
  Interventions: Behavioral: Aerobic training; Behavioral: Cognitive training
- CONTROL group (Experimental): 6-week program of one 20-min session of ROM exercise and one 20-min session of unstructured mental activity 5 days/week.
  Interventions: Behavioral: Range of motion exercise; Behavioral: Unstructured mental activity

INTERVENTIONS:
Behavioral: Aerobic training — One 20-min session of body weight support treadmill training at moderate to high intensity (60-70% heart rate reserve) 5 days/week for 6-weeks.
  Arms: AEROBIC + COGNITIVE group; AEROBIC group
Behavioral: Cognitive training — One 20-min session of cognitive training (computerized dual n-back training program) 5 days/week for 6 weeks.
  Arms: AEROBIC + COGNITIVE group; COGNITIVE group
Behavioral: Range of motion exercise — One 20-min session of range of motion exercise (non-aerobic passive and active movement of upper and lower extremity) 5 days/week for 6-weeks.
  Arms: AEROBIC group; COGNITIVE group; CONTROL group
Behavioral: Unstructured mental activity — One 20-min session of unstructured mental activity (e.g., listening to light novels on tape) 5 days/week for 6-weeks.
  Arms: CONTROL group

SUMMARY:
The objective of the 'Exploring potential synergistic effects of aerobic exercise and cognitive training on cognition after stroke' pilot trial is to investigate the combined effects of aerobic and cognitive training on cognition after stroke. This is to lay the groundwork for a larger RCT on the same topic. Twenty patients greater than 6 months post-stroke will be randomly assigned into one of four following treatment groups: (i) aerobic training (AEROBIC group), (ii) cognitive training (COGNITIVE group), (iii) aerobic exercise plus cognitive training (AEROBIC+COGNITIVE group); and (iv) non-aerobic range of motion (ROM) and unstructured mental activity (CONTROL group) (for group descriptions, please see detailed description below). We hypothesize that the combination of aerobic exercise and cognitive training will be more effective in improving cognition after stroke than either treatment on its own.

DETAILED DESCRIPTION:
Aerobic exercise: Body weight support (BWS) treadmill exercise at moderately high intensity (60-70% of heart rate reserve) using 15-30% BWS. An additional 6-10 min will be needed for warm-up and cool-down. Heart rate will be continuously monitored, and blood pressure and rating of perceived exertion (RPE) will be measured periodically.

Cognitive training: Computerized dual n-back training program that involves a working memory task, the difficulty of which adapts to the individual participant's performance.

ROM exercise: Non-aerobic passive and active movement of upper and lower extremity joints performed with the subject lying on a plinth. RPE will be recorded every 5 minutes to ensure intensity remains low. Mental activities: Unstructured mental activity: such as listening to light novels on tape, which will be selected by the subject from a pre-determined list.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of ischemic or hemorrhagic stroke >6months ago
* Be able to perform a two-step command
* Be able to walk ≥10m with/without aid
* Live within a 75km radius of the QE II
* Pass a cardiology screen for safe participants in exercise training

Exclusion Criteria:

* Have moderate or severe receptive aphasia
* Have terminal illness, life-threatening co-morbidity or concomitant neurological or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-13 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Flanker Test | 10 weeks
  Flanker Test is a computerized test of selective attention and reaction time that involves a motor response. The participant needs to focus and identify an item presented on a screen while ignoring task-irrelevant distractors. Performance on this test has been shown to improve with exercise.
Raven's matrices test | 10 weeks
  A measure of non-verbal reasoning ability and fluid intelligence.
Sternberg digit memory task | 10 weeks
  A measure of visual working memory wherein the subject is shown a set of n digits for study. After a short delay, a digit is shown and the subject is asked to recall whether that item was in the previously viewed set

SECONDARY OUTCOMES:
Peak oxygen consumption | 10 weeks
Fatigue Severity Scale | 10 weeks
  Brief 9-item questionnaire designed to assess patient fatigue
Cognitive Failures Questionnaire | 10 weeks
  A measure of self-reported deficits in completing simple everyday tasks due to failures in attention, memory, perception, and motor function.
Montreal Cognitive Assessment | 10 weeks
Expression of BDNF and IGF-1 in peripheral blood samples | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn MacKay-Lyons, PhD, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia
  - School of Physiotherapy, Dalhousie University, Halifax, Nova Scotia